CLINICAL TRIAL: NCT00618345
Title: Phase II Trial of RAD001 in Relapsed/Refractory Multiple Myeloma
Brief Title: Everolimus in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas E. Witzig, M.D., The Mayo Clinic
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582257; P30CA015083 (NIH); MC048E (Other: Mayo Clinic Cancer Center); 96-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Everolimus; Blotting, Western; Flow Cytometry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: everolimus
Genetic: DNA analysis
Genetic: protein analysis
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response rate in patients with relapsed or refractory multiple myeloma treated with everolimus.

Secondary

* To evaluate the toxicity of everolimus in patients with multiple myeloma.
* To study the tumor cells and blood from patients entering this trial for laboratory correlates.

OUTLINE: Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspirate, biopsy, and blood sample collections periodically. Samples are assessed for the following: cyclin D1, phospho-AKT, phospho-p70 S6 kinase, and phospho-S6 by western blot; checkpoint regulators PTEN, p53, pRB, and p27 by immunoblotting; p53, Rb, p16, PTEN, p27, and cyclin D1 by DNA analysis; caspases 3 and 9 by immunoblotting and Annexin/PI by flow cytometry; unknown molecular markers by protein profiling; and microvessel density.

After completion of study treatment, patients are followed every 3-6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma, meeting 1 of the following criteria:

  * Monoclonal protein in the serum of ≥ 1 g/dL
  * Monoclonal light chain in the urine protein electrophoresis of ≥ 200 mg/24 hours
  * Measurable light chains by free light chain assay of ≥ 10 mg/dL
  * Measurable plasmacytoma
* Must have received prior therapy and have relapsed or refractory disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 2.0 mg/dL (if total bilirubin is elevated, direct bilirubin must be normal)
* AST ≤ 3 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Calcium < 11 mg/dL
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic chemotherapy
* At least 2 weeks since prior biologic therapy or radiotherapy
* At least 2 weeks since prior corticosteroids

  * Concurrent chronic corticosteroids allowed for treatment of disorders other than myeloma
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Confirmed response (complete response, very good partial response, partial response, or minimal response) of serum and urine monoclonal protein

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic; Rafael Fonseca, MD, Principal Investigator — Mayo Clinic; Roy Vivek, MD, Principal Investigator — Mayo Clinic